CLINICAL TRIAL: NCT04396561
Title: Evaluation of Unilateral Ultrasound Guided Paravertebral Block as Perioperative Analgesia For Lower Limb-Sparing Surgery In Adult Cancer Patients: A Prospective, Randomized, Controlled Study
Brief Title: Evaluation of Unilateral Ultrasound Guided Paravertebral Block as Perioperative Analgesia For Lower Limb-Sparing Surgery In Adult Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MS-270-2019
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Unilateral U/S PVB
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled double-blind study.
Who Masked: Participant, Outcomes Assessor
Masking Description: sealed opaque envelopes prepared by an assistant blinded about the study targets and chosen by patient him/herself, allocated into two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Paravertebral group (group P): (Experimental): After induction of general anesthesia and stabilization of the patients, they were positioned in lateral decubitus position with the side to be blocked uppermost.
  Interventions: Drug: Paravertebral group (group P):
- Control group (group C): (Experimental): Patients underwent surgery under general anesthesia and received the perioperative routine protocol of analgesia (IV fentanyl 2 μcg/kg at induction and 1 gm of IV paracetamol).
  Interventions: Drug: Paravertebral group (group P):

INTERVENTIONS:
Drug: Paravertebral group (group P): — In both groups, one reading of mean arterial pressure and heart rate were taken before induction of general anaesthesia and were defined as baseline readings and then were recorded intra-operatively at 15 min intervals.
  Additional bolus doses of fentanyl 0.5µg/kg were given when the mean arterial blood pressure or heart rate raised above 20% of baseline levels.
  Other Names: Control group (group C):

SUMMARY:
Ultrasound imaging has revolutionized the practice of regional anesthesia in that the operator can visualize and identify the paravertebral space, needle during its passage through the tissues, as well as deposition and spread of local anesthetic into the desired spaces. The usage of ultrasound may facilitate more rapid block onset and prolong duration with the added advantage of decrease in drug dosage, reduction in incidence of local anesthetic toxicity, increase success rate, reduction in procedure pain and better patient satisfaction.

DETAILED DESCRIPTION:
Paravertebral block targets drug delivery to the site of pain, thus decreasing opioids use. It can provide greater overall comfort with lower pain scores and greater tolerance of physical activity during the initial postoperative period.

Ultrasound imaging has revolutionized the practice of regional anesthesia in that the operator can visualize and identify the paravertebral space, needle during its passage through the tissues, as well as deposition and spread of local anesthetic into the desired spaces. The usage of ultrasound may facilitate more rapid block onset and prolong duration with the added advantage of decrease in drug dosage, reduction in incidence of local anesthetic toxicity, increase success rate, reduction in procedure pain and better patient satisfaction.

To the best of researchers' knowledge, evaluation of unilateral ultrasound guided paravertebral block as perioperative analgesia for lower limb-sparing surgery in adult cancer patients was not investigated before.

ELIGIBILITY:
Inclusion Criteria:

1. Physical status ASA II and III.
2. Age ≥ 18 and ≤ 65 Years.
3. Body mass index (BMI): > 20 kg/m2 and < 40 kg/m2.
4. Patient undergoing lower limb-sparing surgery for cancer surgeries under general anesthesia.

Exclusion Criteria:

1. Patient refusal.
2. Known sensitivity or contraindication to local anesthetics.
3. History of psychological disorders and/or chronic pain.
4. Coagulopathies with INR ≥1.5: hereditary (e.g. hemophilia, fibrinogen abnormalities & deficiency of factor II) - acquired (e.g. impaired liver functions with PC less than 60 %, vitamin K deficiency & therapeutic anticoagulants drugs).
5. Significant liver or renal insufficiency.
6. Localized infection at the site of block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Total intraoperative fentanyl consumption. | 24 hours
  Total intraoperative fentanyl consumption.

SECONDARY OUTCOMES:
Visual Analouge Scale at 0 , 4 , 8 ,12 ,24 hours postoperatively. | 24 hours
  Visual Analouge Scaleat 0 , 4 , 8 ,12 ,24 hours postoperatively.The VAS consists of a 10-cm line, with anchors at either end. One end is marked "no pain" and the other end is marked "the worst imaginable pain". The patient marks the place on the line to indicate his or her pain intensity. The clinician then measures the line with a ruler and assigns a score.
Heart rate and mean arterial blood pressure . | 24 hours
  Heart rate(beat per minutes) and mean arterial blood pressure(mm HG)
Morphine consumption postoperatively for 24 hours.. | 24 hours Postoperative
  Morphine consumption per mg postoperatively for 24 hours..

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University; Enas Mohamed Samir, M.D, Principal Investigator — Cairo University; Walaa Y Elsabeeny, M.D, Study Director — National Cancer Institute, Cairo University
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Until ending the investigator's work